CLINICAL TRIAL: NCT00608699
Title: A Study to Evaluate the Ability of the HM74A Agonist GSK256073A to Block Niacin-induced Flushing in Healthy Adult Subjects
Brief Title: A Study To See If GSK256073A Can Block Niacin-Induced Flushing In Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: HMA111316
Record Dates: First submitted 2008-01-23; First posted 2008-02-06 (Estimated); Last update posted 2012-04-30 (Estimated); Status verified 2012-04

CONDITIONS: Healthy Subjects; Dyslipidaemias
Keywords: Flushing; GSK256073A,; Dose Escalation,; Immediate Release Niacin,
MeSH Terms: conditions — Flushing

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: GSK256073A tablets + IR niacin tablets — single dosing for 4 to 5 sessions

SUMMARY:
To test the ability of GSK256073 to block niacin-induced flushing when GSK256073 and niacin are co-administered as single doses to HVTs.

ELIGIBILITY:
Inclusion Criteria:

* Adult males between 18 and 55 years of age, inclusive.
* Healthy subjects
* Body weight > 50 kg (110 pounds) and body mass index (BMI) between 19 and 31 where:
* Subjects with QTc < 450 msec at screening

Exclusion Criteria:

* History of significant cardiac arrhythmias
* Active peptic ulcer disease (PUD) and/or history of PUD
* History of gout and/or hyperuricemia
* History of Gilbert's syndrome
* History of recurrent indigestion, stomach upset or diarrhea
* History of other than rare (once yearly or less) flushing
* Recurrent skin rash or psoriasis
* History of kidney stones

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2007-12; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Intensity of reported flushing - visual analogue scale; self reported assessment of flushing | up to 8 hours post dose
Safety and tolerability of GSK256073A and immediate release niacin | up to 36 hours post dose

SECONDARY OUTCOMES:
Standard and Secondary pharmacokinetic endpoints of interest | up to 36 hours post dose
Pharmacodynamic response | up to 36 hours post dose
Pharmacodynamic response | up to 24 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Baltimore, Maryland, United States